CLINICAL TRIAL: NCT00066716
Title: A Phase II Study Of Preoperative Celecoxib/Paclitaxel/Carboplatin For Squamous Cell And Adenocarcinoma Of The Esophagus
Brief Title: Celecoxib, Paclitaxel, and Carboplatin in Treating Patients With Cancer of the Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Nasser Altorki, MD, Weill Cornell Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000316464; NYWCCC-0902-463
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2009-12-08 (Estimated); Status verified 2009-12

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer (lymph node metastasis only)
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Carboplatin; Celecoxib; Paclitaxel; Chemotherapy, Adjuvant; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: carboplatin — Dosed to an AUC of 6 by the Calvert formula, intravenously over 1 hour after paclitaxel on days 1, 22, and 43.
Drug: celecoxib — 400 mg orally BID begins 3-7 days before the first dose of chemotherapy to the morning of surgery. Celecoxib 400 mg orally BID will resume post-operatively 4-8 weeks if there is adequate wound healing and will be continued for 1 year total, that is, 1 year from the date of surgery + 2 weeks unless tumor recurrence is documented.
  Other Names: Celebrex
Drug: paclitaxel — 200 mg/m2 as a 3-hour intravenous infusion on days 1, 22, and 43.
  Other Names: Taxol
Procedure: adjuvant therapy — 1. Surgery will be performed 3-4 weeks after the third dose of paclitaxel and carboplatin.
  2. Operation will be performed within 6-12 hours from the last dose of celecoxib.
  3. Surgery will include an esophagectomy as well as a complete mediastinal and abdominal lymph node dissection.
  4. Celecoxib 400 mg orally BID will resume post-operatively 4-8 weeks if there is adequate wound healing and will be continued for 1 year.
Procedure: conventional surgery — 1. Surgery will be performed 3-4 weeks after the third dose of paclitaxel and carboplatin.
  2. Operation will be performed within 6-12 hours from the last dose of celecoxib.
  3. Surgery will include an esophagectomy as well as a complete mediastinal and abdominal lymph node dissection.
Procedure: neoadjuvant therapy — 1. Surgery will be performed 3-4 weeks after the third dose of paclitaxel and carboplatin.
  2. Operation will be performed within 6-12 hours from the last dose of celecoxib.
  3. Surgery will include an esophagectomy as well as a complete mediastinal and abdominal lymph node dissection.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Celecoxib may increase the effectiveness of a chemotherapy drug by making tumor cells more sensitive to the drug. Celecoxib may also stop the growth of tumor cells by stopping blood flow to the tumor and/or may block the enzymes necessary for their growth. Combining celecoxib with paclitaxel and carboplatin before surgery may shrink the tumor so that it can be removed during surgery. Giving celecoxib alone after surgery may kill any remaining tumor cells.

PURPOSE: This phase II trial is studying how well giving celecoxib together with paclitaxel and carboplatin works in treating patients who are undergoing surgery for esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the rate of complete pathological response and/or minimal residual microscopic disease in patients with squamous cell or adenocarcinoma of the esophagus treated with preoperative celecoxib, paclitaxel, and carboplatin.

Secondary

* Determine the clinical response rate of patients treated with this regimen.
* Determine the chemotherapy-related toxicity of this regimen in these patients.
* Determine the time to progression, disease-free survival, and overall survival of patients treated with this regimen.

OUTLINE: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 1 hour on days 1, 22, and 43. Patients also receive oral celecoxib twice daily beginning 3-7 days before the first dose of chemotherapy and continuing until the morning of planned surgical resection (between days 64 and 71). Approximately 28-56 days after resection, patients may resume oral celecoxib twice daily and continue for 1 year in the absence of disease progression or unacceptable toxicity.

Patients are followed periodically for 18 months after surgery.

PROJECTED ACCRUAL: A total of 39 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed esophageal cancer of 1 of the following cellular types:

  * Squamous cell
  * Adenocarcinoma
* Potentially resectable disease
* No distant metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 80-100%

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* No bleeding disorder

Hepatic

* Bilirubin normal
* AST and ALT less than 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN

Renal

* Creatinine no greater than 2.0 mg/dL

Cardiovascular

* No significant history of unstable cardiovascular disease
* No inadequately controlled hypertension
* No angina
* No myocardial infarction within the past 6 months
* No ventricular cardiac arrhythmias requiring medication
* No congestive heart failure that would preclude study therapy

Pulmonary

* Pulmonary function acceptable for surgery
* No interstitial pneumonia
* No interstitial fibrosis

Gastrointestinal

* No history of peptic ulcer disease
* No irritable bowel syndrome
* No inflammatory bowel disease
* No chronic diarrhea
* No bowel obstruction within the past 5 years

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known hypersensitivity or allergic reactions to COX-2 inhibitors, sulfonamides, NSAIDs, or salicylates
* No hypersensitivity to paclitaxel or carboplatin
* No other serious underlying medical condition that would preclude study therapy
* No significant psychiatric illness that would preclude study compliance
* No uncontrolled diabetes mellitus
* No uncontrolled infection
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* No concurrent chronic steroid use except inhaled mometasone or fluticasone

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 3 weeks since other prior clinical trial therapy
* At least 72 hours since prior nonsteroidal anti-inflammatory drugs (NSAIDs)
* No concurrent chronic NSAID use (7 or more days of continuous therapy per month OR 3 or more days of therapy per week)
* No other concurrent investigational agents
* No concurrent enzyme-inducing anticonvulsants (e.g., phenytoin or phenobarbital)
* No other concurrent cyclo-oxygenase (COX)-2 inhibitors
* No concurrent lithium or fluconazole
* Concurrent low-dose aspirin (325 mg/day or less) allowed for cardiovascular prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2003-06; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Pathological response rate at time of surgical resection | At completion of pathology report.

SECONDARY OUTCOMES:
Clinical response rate | At the time of tumor assessment obtained prior to definitive surgery approximately 1-2 weeks prior to surgical resection.
Disease-free survival | From start of treatment to time of recurrent disease measured postoperatively every 6 months for 18 months.
Overall survival | 18 months after surgery
Toxicities and safety | 30 days after completion of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nasser K. Altorki, MD, Study Chair — Weill Medical College of Cornell University
Locations (1):
- New York Weill Cornell Cancer Center at Cornell University, New York, New York, United States